CLINICAL TRIAL: NCT01590524
Title: Randomized Control Trial for the Effect of Guided Imagery and Progressive Muscle Relaxation in Reducing Anxiety for Parents of Hospitalized Children With Cancer
Brief Title: Feasibility Study on the Effect of Complementary Methods as Supportive Interventions for Parents of Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, Dr. Andreas Charalambous, Lecturer-Researcher, Cyprus University of Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: AC-GIPMRL-87
Record Dates: First submitted 2012-02-08; First posted 2012-05-03 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Anxiety; Stress; Mood; Coping
Keywords: Parent; childhood cancer; Complementary and Alternative
MeSH Terms: conditions — Anxiety Disorders; Neoplasms | interventions — Imagery, Psychotherapy; Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAM group (Experimental): Subjects receiving the interventions and standard psychological care
  Interventions: Behavioral: Guided Imagery and Progressive Muscle Relaxation
- No-CAM group (No Intervention): Parents receiving only standard psychological care

INTERVENTIONS:
Behavioral: Guided Imagery and Progressive Muscle Relaxation — Daily implementation of the guided imagery and progressive muscle relaxation techniques additionally to weekly supervised sessions.
  Arms: CAM group

SUMMARY:
The purpose of this study is to determine whether Guided Imagery and Progressive Muscle relaxation are effective as stress reducing techniques in parents of hospitalized children with cancer.

DETAILED DESCRIPTION:
Having a children with cancer can be a source of stress for parents during hospitalization. The stress experienced by the parents can negatively influence their functionality, daily activities, psychological state and also their physical condition. The studies in the literature have mainly focused on the child rather than the parent, and studies specifically for guided imagery are scarce. Since the parents are often neglected by the healthcare professionals during the stress evoking period of hospitalization, this study will test the effectiveness of complementary methods in improving the psychological state of the parents.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate
* having a child with childhood cancer been hospitalized for 4 weeks
* have a child (0-18) of age with childhood cancer
* able to speak and write Greek fluently
* no previous experience with CAM techniques

Exclusion Criteria:

* receiving drug therapy for stress
* using another CAM technique during the study

  * parents of children receiving palliative care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Changes in the number of Participants with anxiety | 1 week, 2 week, 3 week , 4 week
  Participants response to the complementary and alternative intervention will be measured through their scores on the Hamilton Anxiety Scale

SECONDARY OUTCOMES:
Changes in the number of Participants with mood changes | 1 week, 2 week, 3 week , 4 week
  Participants response to the complementary and alternative interventions will be measured through their scores on the POMS scale
stress level with Biodots | 1 week, 2 week, 3 week, 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Charalambous, PhD, Principal Investigator — Cyprus University of Technology
Locations (1):
- Archbishob Makarios Hospital, Nicosia, Nicosia, Cyprus